CLINICAL TRIAL: NCT05047354
Title: Natural History Investigation Into Biochemical and Phenotypical Aspects of Smith-Lemli-Opitz Syndrome and Related Disorders of Cholesterol Metabolism
Brief Title: Biochemical and Phenotypical Aspects of Smith-Lemli-Opitz Syndrome and Related Disorders of Cholesterol Metabolism
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000487; 000487-CH
Record Dates: First submitted 2021-09-16; First posted 2021-09-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Smith Lemli Opitz Syndrome; CHILD Syndrome; Lathosterolosis; Desmosterolosis
Keywords: 7-dehydrocholesterol reductase; 7-dehydrocholesterol; cholesterol deficiency; Natural History
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome; Congenital Hemidysplasia with Ichthyosiform Erythroderma and Limb Defects; Lathosterolosis; Desmosterolosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Subjects with Smith-Lemli-Opitz syndrome
- 2: Subjects with Disorders of cholesterol synthesis and metabolism

SUMMARY:
Background:

Smith-Lemli-Opitz Syndrome (SLOS) is a genetic disorder. It can cause birth defects and developmental delays. There is no cure for SLOS or other inherited diseases related to cholesterol production or storage. The data gained in this study may help researchers find ways to measure how well future treatments work.

Objective:

To learn more about SLOS and related disorders and how these diseases affect participants and relatives.

Eligibility:

People of any age who have or are suspected to have SLOS or another inherited disease related to cholesterol production or storage. Relatives are also needed.

Design:

Participants will be screened with a medical record review.

Participants will have visits every 6 to 12 months. They will have a physical exam. They will fill out a survey about their medical and behavioral history. They may have an eye exam. They may have a neurodevelopmental assessment. They may have a hearing test. Their outer and middle ears may be examined. Their ability to speak, understand speech, eat, and swallow may be assessed. They may get X-rays while they chew and swallow. Their functional ability and needs for adaptive devices or braces may be assessed. They may have a lumbar puncture. Photographs may be taken of their face and body.

Participants who cannot visit the NIH and relatives will have a virtual visit once a year. They will talk about their medical history and symptoms. They give blood, urine, and skin samples at a lab near their home. They will fill out a survey about their medical and behavioral history.

Participation will last for several years.

DETAILED DESCRIPTION:
Study Description: The objective of this study is to characterize the natural history of Smith-Lemli-Opitz Syndrome (SLOS) and related disorders (such as lathosterolosis, desmosterolosis, X-linked dominant chondrodysplasia punctata (CDPX2), CHILD syndrome, HEM dysplasia, and Antley-Bixler syndrome) by collecting both crosssectional and longitudinal data on individuals with these conditions.

Our goal is to investigate genetic, biochemical, and clinical aspects of SLOS and related disorders in order to facilitate development and implementation of future therapeutic trials. This protocol consists of a main study and three sub-studies. The main study involves inperson evaluation of patients and carriers of SLOS and related disorders. The first sub-study includes collecting biorepository samples from patients and carriers of SLOS and related disorders. The second sub-study involves obtaining a telemedicine history and full review of systems for affected individuals with SLOS and related disorders. The third sub-study involves a survey of caregivers of

deceased individuals with SLOS, which will address questions regarding the deceased individual s medical history and inform causes of death. All questions in the survey will be regarding the deceased individual s medical history, none of the questions will be about the caregivers. This protocol will also maintain a database of information collected over the past two decades at the NIH on SLOS trial participants. All individuals with SLOS, related disorders and carriers will be eligible for enrollment.

Objectives: The primary objective of this study is to determine laboratory or clinical outcome measures that could be used in future therapeutic trials.

The secondary objectives of these studies are to define comorbidities and mortality of the disease, investigate the causes of mortality, identify potential participants for future therapeutic trials and evaluate possible laboratory outcome measures and biomarkers in carriers and suspected carriers.

Endpoints: Primary endpoints

1. Phenotypic characterization of individuals with SLOS and related inborn errors of cholesterol synthesis. Define and characterize disease related morbidity and mortality.
2. Establishing a biomaterial collection (Blood, urine, CSF, DNA/RNA and cell lines) corresponding to well-phenotyped individuals for biomarker discovery and characterization.

Secondary endpoints: Phenotypic history as well as blood and urine biomarkers in individuals heterozygous for pathogenic DHCR7 variants or pathogenic variants in cholesterol synthetic genes. Additional outcomes include assessments of bone health.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females of any age with any one of the following:

* Clinical, biochemical, or genetic diagnosis of Smith-Lemli-Opitz Syndrome OR
* Clinical, biochemical, or genetic diagnosis of desmosterolosis, lathosterolosis, CHILD syndrome, X-linked dominant chondrodysplasia type2 or another inborn error of cholesterol synthesis OR
* Clinical suspicion of an inborn error of cholesterol synthesis, metabolism or impaired cholesterol homeostasis. Clinical observations may include, but are not limited to lipid-laden macrophages, abnormal LDL, HDL, total cholesterol, triglycerides, abnormal lipid

electrophoresis, lipid storage in other tissues. OR

-Biologic parents of affected individuals or known carriers based on previously done genetic testing who are willing and able to provide samples of any or all of the following: blood, urine, a skin biopsy, and/or tissue derived from clinically indicated surgery or autopsy.

EXCLUSION CRITERIA:

* Affected individuals who cannot travel to the NIH because of their medical condition will be excluded from on-site participation. They may participate in the telemedicine or in the biomaterials parts of the study.
* Affected individuals who, in the opinion of the investigator, are unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation will be excluded from on-site participation. They may participate in the telemedicine or in the

biomaterials parts of the study.

* Carrier adults who are unable to or unwilling to provide any of the following samples: Blood, urine, skin biopsy sample or tissue derived from clinically indicated surgery or skin biopsy.
* Female participants who are pregnant will be excluded from evaluations requiring sedation, radiation and LP. Total blood draw volumes will be kept at a minimum or if anemia of pregnancy is known, no blood will be taken for research testing.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or female of any age with disorder of cholesterol metabolism. No geographic restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2031-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine laboratory or clinical outcome measures that could be used in future therapeutic trials. | ongoing
  We will obtain data from patient evaluations that may be used as therapeutic targets in the fututre.
The secondary objectives of these studies are to define comorbidities and mortality of the disease, to identify potential participants for future therapeutic trials and to evaluate possible laboratory outcome measures in carriers and suspected c... | ongoing
  To describe in more detail long term manifestations of SLOS and disorders of cholesterol synthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nowaczyk MJ, Irons MB. Smith-Lemli-Opitz syndrome: phenotype, natural history, and epidemiology. Am J Med Genet C Semin Med Genet. 2012 Nov 15;160C(4):250-62. doi: 10.1002/ajmg.c.31343. Epub 2012 Oct 11. PMID 23059950
- [Background] Irons M, Elias ER, Salen G, Tint GS, Batta AK. Defective cholesterol biosynthesis in Smith-Lemli-Opitz syndrome. Lancet. 1993 May 29;341(8857):1414. doi: 10.1016/0140-6736(93)90983-n. No abstract available. PMID 7684480
- [Background] SMITH DW, LEMLI L, OPITZ JM. A NEWLY RECOGNIZED SYNDROME OF MULTIPLE CONGENITAL ANOMALIES. J Pediatr. 1964 Feb;64:210-7. doi: 10.1016/s0022-3476(64)80264-x. No abstract available. PMID 14119520
- [Derived] Selvaraman A, Rahhal S, Bianconi S, Furnary T, Porter FD. Assessing Postnatal Mortality in Smith-Lemli-Opitz Syndrome. Am J Med Genet A. 2025 Feb;197(2):e63875. doi: 10.1002/ajmg.a.63875. Epub 2024 Sep 13. PMID 39271956
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000487-CH.html